CLINICAL TRIAL: NCT02594696
Title: Proactive Psychiatry Consultation for Patients With Cancer and Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kelly Edwards Irwin, Instructor, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-293; 5R25CA092203-13 (NIH)
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Major Depression; Schizophrenia; Bipolar Disorder; Lung Cancer; Breast Cancer; Head and Neck Cancer; GI Cancer; Cancer
Keywords: Major depression and Cancer; Schizophrenia and Cancer; Bipolar disorder and Cancer; Lung Cancer; Breast Cancer; Head and Neck cancer; GI cancer; Schizophrenia; Bipolar disorder
MeSH Terms: conditions — Depressive Disorder, Major; Schizophrenia; Bipolar Disorder; Lung Neoplasms; Breast Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proactive Psychiatry Consultation (PPC) (Experimental): The patient is linked to a psychiatrist and case manager at cancer diagnosis who deliver team-based, patient-centered care. The psychiatrist collaborates with the oncologist to guide cancer treatment. The psychiatrist and case manager proactively monitor patient symptoms and potential barriers to care and remain in communication with the patient, oncology team, and community-based providers for the duration of the intervention.
  * Patients complete study assessments at baseline, 4 +/- 2 weeks after baseline, and post-intervention (12 +/-2 weeks after baseline)
  * Oncologists provide feedback about the usefulness of the intervention (12 +/- 2 weeks after baseline)
  Interventions: Other: Proactive Psychiatry Consultation (PPC)

INTERVENTIONS:
Other: Proactive Psychiatry Consultation (PPC) — * The psychiatrist conducts a tailored, cancer-specific assessment to optimize psychiatric symptoms and collaborates with the oncologist to develop and modify the cancer treatment plan.
  * The case manager, a social worker, engages with the patient to promote self-management, identify and address barriers to care, and bridge communication with oncology and mental health.
  * The psychiatrist and case manager proactively monitor symptoms and the process of cancer care, remain in regular contact with the patient and communicate with the oncology team at least every 4 weeks
  * The psychiatrist and case manager are available for consultation across care settings (outpatient, inpatient, home).
  * Recommendations are documented in the medical record and communicated directly to the oncology team

SUMMARY:
Individuals with severe mental illness (SMI) including schizophrenia and bipolar disorder are dying younger than the general population; cancer is a leading cause of death in this population. People with SMI have higher rates of dying from breast, lung, and colon cancer, and disparities in treatment appear to be one contributing factor. Individuals with SMI may be diagnosed with more advanced stage cancer and less likely to receive stage-appropriate cancer treatment. Although collaborative care models integrating medical and psychiatric care have shown promise in other populations, the challenge of treating SMI and cancer is distinct and relatively understudied. Patients may have uncontrolled psychiatric symptoms that can impact their understanding of their diagnosis and treatment decisions. Oncologists have less training and inadequate time to address multiple unmet needs. Mental health care is frequently fragmented from cancer care.

The investigators want to understand if it is helpful for patients with SMI to be connected to a psychiatrist and case manager when cancer is diagnosed. Optimizing psychiatric symptoms and facilitating communication between the patient, the oncology team, and mental health providers may improve care. The goal is to pilot a pragmatic intervention for patients with cancer and SMI that can be integrated into cancer care, is acceptable to patients and oncology clinicians, and may promote the delivery of stage-appropriate cancer treatment to an underserved population.

Patients will be connected to a psychiatrist and case manager at cancer diagnosis who will follow the patient and communicate with the oncology team during the 12 week intervention. All participants will complete brief surveys at baseline, 4 weeks, and 12 weeks. Oncology clinicians will provide feedback about the intervention at 12 weeks. Cancer treatment received and healthcare utilization will be assessed at 6 months post-intervention.

DETAILED DESCRIPTION:
Specific Aims:

Aim 1: To evaluate the feasibility and acceptability of proactive psychiatry consultation and case management among individuals with SMI treated at the MGH Cancer Center and their oncology clinicians.

Aim 2: To describe the rates of receipt of stage-appropriate cancer treatment and patterns of healthcare utilization in patients with SMI and cancer who are receiving the intervention

Aim 3: To explore patterns of change in psychiatric symptoms, quality of life, illness understanding, and alliance with the oncology clinician in patients with SMI and a recent cancer diagnosis who are receiving the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of a primary psychotic disorder (schizophrenia, schizoaffective disorder, delusional disorder), bipolar disorder, or major depressive disorder with prior psychiatric hospitalization, confirmed by diagnostic assessment of the PI, a psychiatrist with expertise in SMI and cancer
* Within 8 weeks of initial oncology consultation at the MGH Cancer Center (patients who come for a second opinion and opt to have their cancer treatment at MGH will be considered eligible, patients who have been treated previously for other types of cancer will be considered eligible).
* Age >18 years old, verbal fluency in English
* Suspected or newly diagnosed lung, GI, head/neck, or breast cancer documented in initial oncology note or confirmed by pathology

Exclusion Criteria:

* Cognitive impairment severe enough to interfere with completing the study assessments or providing informed consent
* History of dementia or traumatic brain injury
* Refuse participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing the intervention in patients with SMI and cancer | 12 weeks
  Feasibility of participating in the intervention:
  * At least 75% of intervention participants complete the psychiatric diagnostic assessment and establish contact with the case manager
  * At least 75% of enrolled patients complete the patient-reported measures.
  Feasibility of enrollment process:
  • At least 50% of patients who are approached enroll in the intervention

SECONDARY OUTCOMES:
Acceptability of the intervention for patients with SMI and cancer and oncology clinicians | 12 weeks
  Study acceptability will be evaluated via exit interviews with oncology clinicians and study participants regarding the content, timing, and usefulness of the intervention.
Rates of receipt of stage-appropriate cancer treatment | 6 Months
  Rates of receipt of stage-appropriate cancer treatment measured by medical record review and feedback from oncology clinician at 6 months post intervention
Rates of receipt of healthcare utilization in the outpatient setting | 6 Months
  Rates of healthcare utilization in outpatient setting measured by medical record review at 6 months post intervention
Rates of receipt of healthcare utilization in the acute care setting | 6 Months
  Rates of healthcare utilization in acute care setting (aggregate measure of emergency visits and hospitalizations) measured by medical record review at 6 months post intervention
Change in clinician-rated psychiatric symptoms | Baseline to 12 weeks post intervention
  - Psychiatric symptom severity according to the Behavioral Psychiatric Rating Scale (BPRS) pre and 12 weeks post intervention
Change in clinician-rated psychiatric illness severity | Baseline to 12 weeks post intervention
  - Psychiatric illness severity according to the Clinical Global Impression-Severity (CGI-S) scale pre-intervention, 4 weeks post intervention, and 12 weeks post intervention
Change in self-reported psychiatric symptoms | Baseline to 12 weeks post intervention
  - Self reported psychiatric symptoms according to the Behavior and Symptoms Identification Scale (BASIS) pre, 4 weeks post intervention, and 12 weeks post intervention
Change in self-reported depression symptoms | Baseline to 12 weeks post intervention
  - Self-reported severity of depression according to the Patient Health Questionnaire-9 (PHQ-9) pre, 4 weeks post-intervention, and 12 weeks post-intervention
Change in quality of life | Baseline to 12 weeks post intervention
  -Quality of life according to the Functional Assessment of Cancer Therapy-General (FACT-G)pre, 4 weeks post intervention, and 12 weeks post intervention
Change in illness understanding | Baseline to 12 weeks post intervention
  Self-reported illness understanding according to the Prognosis and Treatment Perceptions Questionnaire at baseline and 12 weeks post intervention
Change in alliance with the oncology clinician | Baseline to 12 weeks post intervention
  Self-reported alliance with the oncology clinician according to the Human Connection Scale at baseline and 12 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Irwin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States